CLINICAL TRIAL: NCT00961935
Title: Examining Neurocognitive Profiles of Bipolar Disorder and Attention-Deficit Hyperactivity Disorder
Brief Title: Pediatric Bipolar Disorder Study at UCLA
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); The State Family Fund (Unknown)
Responsible Party: Principal Investigator, James McCracken, Chair, University of California, Los Angeles
Other Study IDs: P50MH077248-02 (NIH); P50MH077248-02 (NIH); DNBBS B2-MBP (Other Grant/Funding Number: National Institute of Mental Health)
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; child bipolar disorder; adolescent bipolar disorder; pediatric bipolar disorder; fMRI; MRI; EEG; neurocognitive tasks
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The UCLA Semel Institute for Neuroscience in Los Angeles, CA, is conducting a study looking at similarities and differences in how the brain works between bipolar disorder and attention deficit hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
Children between the ages of 7 and 17 years old, with a diagnosis of Bipolar I, Bipolar II, or Bipolar NOS, are currently being recruited for this study looking at similarities and differences in how the brain works between bipolar disorder and attention deficit hyperactivity disorder (ADHD). The study involves a comprehensive evaluation at intake, cognitive assessment, EEG, and functional MRI, done over the course of 2 or 3 visits. This study does not provide treatment. However, with participants' consent, the assessment information can be shared with the child's clinician or psychiatrist and a letter with the results from cognitive testing can be prepared, which can be useful in school planning. Referrals for treatment can also be provided.

ELIGIBILITY:
Inclusion Criteria:

* Subject suffers clinically impairing symptoms of mood lability.
* Child has resided with primary caretaker for at least 6 months.
* Caretaker speaks sufficient English to complete all study evaluations and measures.

Exclusion Criteria:

* Lifetime history of mental retardation, autism, or primary diagnosis of psychosis.
* Subject is pregnant or nursing.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Bipolar Disorder
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-08; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Walshaw, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute for Neuroscience and Human Behavior, Los Angeles, California, United States

REFERENCES:
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Bearden CE, Hoffman KM, Cannon TD. The neuropsychology and neuroanatomy of bipolar affective disorder: a critical review. Bipolar Disord. 2001 Jun;3(3):106-50; discussion 151-3. doi: 10.1034/j.1399-5618.2001.030302.x. PMID 11465675
- [Background] Blumberg HP, Leung HC, Skudlarski P, Lacadie CM, Fredericks CA, Harris BC, Charney DS, Gore JC, Krystal JH, Peterson BS. A functional magnetic resonance imaging study of bipolar disorder: state- and trait-related dysfunction in ventral prefrontal cortices. Arch Gen Psychiatry. 2003 Jun;60(6):601-9. doi: 10.1001/archpsyc.60.6.601. PMID 12796223
- [Background] Carlson GA. Mania and ADHD: comorbidity or confusion. J Affect Disord. 1998 Nov;51(2):177-87. doi: 10.1016/s0165-0327(98)00179-7. PMID 10743850
- [Background] Carlson GA. Juvenile mania versus ADHD. J Am Acad Child Adolesc Psychiatry. 1999 Apr;38(4):353-4. doi: 10.1097/00004583-199904000-00001. No abstract available. PMID 10199100
- [Background] Casey BJ, Castellanos FX, Giedd JN, Marsh WL, Hamburger SD, Schubert AB, Vauss YC, Vaituzis AC, Dickstein DP, Sarfatti SE, Rapoport JL. Implication of right frontostriatal circuitry in response inhibition and attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 1997 Mar;36(3):374-83. doi: 10.1097/00004583-199703000-00016. PMID 9055518
- [Background] Castellanos FX, Giedd JN, Eckburg P, Marsh WL, Vaituzis AC, Kaysen D, Hamburger SD, Rapoport JL. Quantitative morphology of the caudate nucleus in attention deficit hyperactivity disorder. Am J Psychiatry. 1994 Dec;151(12):1791-6. doi: 10.1176/ajp.151.12.1791. PMID 7977887
- [Background] Faraone SV, Biederman J, Wozniak J, Mundy E, Mennin D, O'Donnell D. Is comorbidity with ADHD a marker for juvenile-onset mania? J Am Acad Child Adolesc Psychiatry. 1997 Aug;36(8):1046-55. doi: 10.1097/00004583-199708000-00012. PMID 9256584
- [Background] Geller B, Luby J. Child and adolescent bipolar disorder: a review of the past 10 years. J Am Acad Child Adolesc Psychiatry. 1997 Sep;36(9):1168-76. doi: 10.1097/00004583-199709000-00008. PMID 9291717
- [Background] Geller B, Tillman R, Craney JL, Bolhofner K. Four-year prospective outcome and natural history of mania in children with a prepubertal and early adolescent bipolar disorder phenotype. Arch Gen Psychiatry. 2004 May;61(5):459-67. doi: 10.1001/archpsyc.61.5.459. PMID 15123490
- [Background] Geller B, Williams M, Zimerman B, Frazier J, Beringer L, Warner KL. Prepubertal and early adolescent bipolarity differentiate from ADHD by manic symptoms, grandiose delusions, ultra-rapid or ultradian cycling. J Affect Disord. 1998 Nov;51(2):81-91. doi: 10.1016/s0165-0327(98)00175-x. PMID 10743841
- [Background] Geller B, Zimerman B, Williams M, Delbello MP, Bolhofner K, Craney JL, Frazier J, Beringer L, Nickelsburg MJ. DSM-IV mania symptoms in a prepubertal and early adolescent bipolar disorder phenotype compared to attention-deficit hyperactive and normal controls. J Child Adolesc Psychopharmacol. 2002 Spring;12(1):11-25. doi: 10.1089/10445460252943533. PMID 12014591
- [Background] Gruber SA, Rogowska J, Yurgelun-Todd DA. Decreased activation of the anterior cingulate in bipolar patients: an fMRI study. J Affect Disord. 2004 Oct 15;82(2):191-201. doi: 10.1016/j.jad.2003.10.010. PMID 15488247
- [Background] Kaufman J, Birmaher B, Brent D, Rao U, Flynn C, Moreci P, Williamson D, Ryan N. Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL): initial reliability and validity data. J Am Acad Child Adolesc Psychiatry. 1997 Jul;36(7):980-8. doi: 10.1097/00004583-199707000-00021. PMID 9204677
- [Background] Kent L, Craddock N. Is there a relationship between attention deficit hyperactivity disorder and bipolar disorder? J Affect Disord. 2003 Feb;73(3):211-21. doi: 10.1016/s0165-0327(02)00092-7. PMID 12547289
- [Background] Kovatchev B, Cox D, Hill R, Reeve R, Robeva R, Loboschefski T. A psychophysiological marker of attention deficit/hyperactivity disorder (ADHD)--defining the EEG consistency index. Appl Psychophysiol Biofeedback. 2001 Jun;26(2):127-40. doi: 10.1023/a:1011339206875. PMID 11480163
- [Background] Mostofsky SH, Cooper KL, Kates WR, Denckla MB, Kaufmann WE. Smaller prefrontal and premotor volumes in boys with attention-deficit/hyperactivity disorder. Biol Psychiatry. 2002 Oct 15;52(8):785-94. doi: 10.1016/s0006-3223(02)01412-9. PMID 12372650
- [Background] National Institute of Mental Health research roundtable on prepubertal bipolar disorder. J Am Acad Child Adolesc Psychiatry. 2001 Aug;40(8):871-8. doi: 10.1097/00004583-200108000-00007. PMID 11501685
- [Background] Quraishi S, Frangou S. Neuropsychology of bipolar disorder: a review. J Affect Disord. 2002 Dec;72(3):209-26. doi: 10.1016/s0165-0327(02)00091-5. PMID 12450638
- [Background] Pennington BF, Ozonoff S. Executive functions and developmental psychopathology. J Child Psychol Psychiatry. 1996 Jan;37(1):51-87. doi: 10.1111/j.1469-7610.1996.tb01380.x. PMID 8655658
- [Background] Sax KW, Strakowski SM, Zimmerman ME, DelBello MP, Keck PE Jr, Hawkins JM. Frontosubcortical neuroanatomy and the continuous performance test in mania. Am J Psychiatry. 1999 Jan;156(1):139-41. doi: 10.1176/ajp.156.1.139. PMID 9892312
- [Background] Walcott CM, Landau S. The relation between disinhibition and emotion regulation in boys with attention deficit hyperactivity disorder. J Clin Child Adolesc Psychol. 2004 Dec;33(4):772-82. doi: 10.1207/s15374424jccp3304_12. PMID 15498744
- [Background] Wilder-Willis KE, Sax KW, Rosenberg HL, Fleck DE, Shear PK, Strakowski SM. Persistent attentional dysfunction in remitted bipolar disorder. Bipolar Disord. 2001 Apr;3(2):58-62. doi: 10.1034/j.1399-5618.2001.030202.x. PMID 11333063
- [Background] Wozniak J, Biederman J, Kiely K, Ablon JS, Faraone SV, Mundy E, Mennin D. Mania-like symptoms suggestive of childhood-onset bipolar disorder in clinically referred children. J Am Acad Child Adolesc Psychiatry. 1995 Jul;34(7):867-76. doi: 10.1097/00004583-199507000-00010. PMID 7649957